CLINICAL TRIAL: NCT01116518
Title: Treatment of Atraumatic Rotator Cuff Rupture in Elderly Patients
Acronym: toarcriep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Tampere University Hospital (Other); Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Ville Aarimaa, Ville Äärimaa, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 106/2007
Record Dates: First submitted 2010-04-29; First posted 2010-05-05 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2010-05

CONDITIONS: Atraumatic Rotator Cuff Rupture
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- physiotherapy (Active Comparator)
  Interventions: Procedure: physiotherapy
- acromioplasty (Active Comparator)
  Interventions: Procedure: acromioplasty
- acromioplasty and rotator cuff reconstruction (Active Comparator)
  Interventions: Procedure: acromioplasty and rotator cuff reconstruction

INTERVENTIONS:
Procedure: physiotherapy
  Arms: physiotherapy
Procedure: acromioplasty
  Arms: acromioplasty
Procedure: acromioplasty and rotator cuff reconstruction
  Arms: acromioplasty and rotator cuff reconstruction

SUMMARY:
The purpose of the investigators study is to compare the effect of: 1) physiotherapy 2) arthroscopic acromioplasty and debridement or 3) arthroscopic rotator cuff reconstruction and acromioplasty in the treatment of degenerative, atraumatic rotator cuff rupture.

DETAILED DESCRIPTION:
The study will be conducted according to the revised Declaration of Helsinki by The World Medical Association and the ICH-guidelines for good clinical trial practice. The study will be submitted for approval to the Ethics Committee of the Hospital District of Varsinais-Suomi, Finland. A written informed consent will be obtained from each patient.

This study will be conducted at three different hospitals i.e. Turku University Hospital, Tampere University Hospital (Hatanpää hospital) and Kuopio University Hospital as a multicenter study. A total of 180 patients, 60 patients at each hospital, will be included in this study. The patients are clinically examined and a routine x-ray and MRI-investigation are performed. Patients must have an atraumatic degenerative supraspinatus tendon rupture comprising less than 2/3 of the tendon insertion, i.e. 1/3 of the tendon insertion must be intact. The rupture must be documented by MRI investigation. Patients must be willing and give a written informed consent. After recruitment the patients are randomized in one of three studied treatment modalities. The randomization is made after clinical and MRI investigation by neutral attendant using sealed envelopes. 60 identical envelopes (20 per group) are made in each center.

The Constant score is used as a primary outcome measure. The Constant score is measured from each patient right before treatment intervention and at three and six months, one, two and five years after the intervention. The intervention groups are designed in a cumulative fashion: structured and standardized physiotherapy treatment proceeds gradually in all patients (groups 1,2,3), in addition to physiotherapy patients in group 2 are treated with acromioplasty, and patients in group 3 with acromioplasty and rotator cuff reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. age over 55 years
2. atraumatic penetrating supraspinatus tendon rupture comprising less than 2/3 of the tendon insertion and documented with MRI investigation.
3. full active range of motion
4. written informed consent from participating subject

Exclusion Criteria:

1. age under 55 years
2. existing significant malignant, haematological, endocrine, metabolic, rheumatoid or gastrointestinal disease
3. cytostatic or corticosteroid medication
4. glenohumeral osteoarthrosis grade III or above (X-ray evaluation with present osteophytes according to Kellgren-Lawrence classification)
5. history of alcoholism, drug abuse, psychological or other emotional problems that are likely to invalidate informed consent
6. previous same shoulder surgery
7. a massive tendon tear involving the whole supraspinatus tendon and/or combined tear of two - three tendons ie. supraspinatus with infraspinatus or subscapularis tendon tear.
8. patients denial

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Shoulder score by Constant and Murley | 2 years
  Constant scoring is endorsed by SECEC/ESSSE and is the most largely used instrument measuring shoulder pain, function and strenght. This scoring system is very suited for evaluating disability caused by rotator cuff ruptures.
Constant score
  subjective and objective shoulder score

CONTACTS AND LOCATIONS:
Overall Officials: Juha Kukkonen, MD, Principal Investigator — Turku University Hospital; Ville Äärimaa, MD, PhD, Study Director — Turku University Hospital
Locations (3):
- Finland (3):
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku